CLINICAL TRIAL: NCT04262557
Title: Evaluation of the Correlation Between the Respiratory Index Events Generated by Sunrise® Versus Polysomnography for Sleep Apnea Syndrome Diagnosis
Brief Title: Sunrise® a New Medical Device to Diagnose Sleep Apnea Syndrome
Acronym: SENSAPNEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Sunrise (Industry); Icadom (Industry); DOCAPOST (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC19.358
Record Dates: First submitted 2020-02-04; First posted 2020-02-10 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Sleep Apnea Syndrome, Obstructive
Keywords: New medical device; Mandibular movement; Respiratory event index; Polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Polysomnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sunrise+PSG (Experimental): PSG and Sunrise® will be set at the patient's home by IC@dom. The first night, the patient will be equipped by both PSG and Sunrise® and only by the Sunrise® for the two following nights.
  Interventions: Diagnostic Test: Sunrise® solution; Diagnostic Test: Polysomnography

INTERVENTIONS:
Diagnostic Test: Sunrise® solution — Type II medical device with the CE label. It is a chin sensor associated to an integrated and connected platform.
Diagnostic Test: Polysomnography — Gold standard method to diagnose SAS used as comparator
  Other Names: PSG

SUMMARY:
Sleep Apnea Syndrome (SAS) is a serious health issue that should be managed in order to limit its adverse health consequences. SAS is known to induce cardiovascular diseases, diabetes and depression. The prevalence of SAS is still growing with social and economic repercussion. Today, polysomnography (PSG) is the gold standard reference method for SAS diagnosis. However, it is a constraining and expensive technology. In order to improve patients' life quality, many new technologies have been developed for the SAS diagnosis.

The aim of this study is to evaluate the Sunrise®, a new medical integrated solution for SAS diagnosis, in comparison with PSG. This solution consists in a chin sensor recording mandibular movements and measuring the respiratory event index (ERI) through an artificial intelligence algorithm analysis.

DETAILED DESCRIPTION:
Sunrise® is a type IIa medical device with the CE label. It is a new home sleep technology, non-invasive, reliable and affordable by the patient.

The objective of this study is to evaluate the efficiency of the device in comparison with PSG for sleep apnea diagnosis.

40 subjects, suspected to be apneic, will be equipped at home by the chin sensor, the Sunrise® device, recording their mandibular movements while sleeping. The Sunrise® solution will provide the respiratory event index (REI) as well as the respiratory micro-arousals.

Inclusion visit will be executed at the University Hospital Grenoble Alpes. However, PSG and Sunrise® will be set at the patient's home by IC@dom. The first night, the patient will be equipped by both PSG and Sunrise® and only by the Sunrise® for the two following nights.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected to have a sleep apnea syndrome (Berlin score≥2)
* Able to use a smartphone application
* Be legally able to give consent
* Person affiliated to social security

Exclusion Criteria:

* Patients already treated for SAS
* Patients suffering from a chronic obstructive or restrictive pulmonary disease with or without oxygen.
* Patients suffering from a unstable cardiovascular disease or a severe heart failure requiring an hospitalzation in the previous three months or conform with the New York Heart Association criteria for class II or III diseases
* Patients treated with myorelaxant medicines
* Patients with a long beard disabling the setting of the mandibular sensor
* Subjects listed in articles L1121-5 à L1121-8: Pregnant women, feeding and parturient; subject under administrative or judicial control, persons who are protected under the act.
* Person in exclusion period for another study or participating in a medical study testing drugs.
* Subjects not being cooperative or respecting the study instructions, according the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
The performance of Sunrise® to detect the respiratory event index (REI) | 1 night
  Evaluation of the correlation between Sunrise® and PSG for the estimation of the REI

SECONDARY OUTCOMES:
Evaluation of the Sunrise® reproductibility on three consecutive nights | 3 nights
  REI measured by Sunrise® on three consecutive nights
Evaluation of the sleep quality: depth of sleep | 3 nights
  Depth of sleep was assessed by the St Mary Hospital Questionnaire Q1 (scale from 1 "very light" to 8 "very depth"), after one night without device, one night with PSG+Sunrise® and one night with Sunrise® only
Evaluation of the sleep quality: number of wake-ups | 3 nights
  Number of Wake-ups was assessed by the St Mary Hospital Questionnaire Q2 (scale from 0 "no Wake-up" to 7 "more than 6 Wake-ups"), after one night without device, one night with PSG+Sunrise® and one night with Sunrise® only
Evaluation of the sleep quality: sleep duration | 3 nights
  Sleep duration was assessed by the St Mary Hospital Questionnaire Q3 (in hour), after one night without device, one night with PSG+Sunrise® and one night with Sunrise® only

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis Pépin, MD, PhD, Principal Investigator — University Hospital Grenoble Alpes
Locations (1):
- University Hospital Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kelly JL, Ben Messaoud R, Joyeux-Faure M, Terrail R, Tamisier R, Martinot JB, Le-Dong NN, Morrell MJ, Pepin JL. Diagnosis of Sleep Apnoea Using a Mandibular Monitor and Machine Learning Analysis: One-Night Agreement Compared to in-Home Polysomnography. Front Neurosci. 2022 Mar 15;16:726880. doi: 10.3389/fnins.2022.726880. eCollection 2022. PMID 35368281